CLINICAL TRIAL: NCT02875964
Title: Definition of Links Between Non-invasives Methods and Intracerebral EEG With Simultaneous Recordings.
Acronym: MEG-SEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-16; 2012-A00644-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography; Magnetoencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- registration of intracerebral activity (Experimental): epileptic patient receiving implantation of intracranial electrodes
  Interventions: Device: electroencephalogram; Device: magnetoencephalogram

INTERVENTIONS:
Device: electroencephalogram — Implanting electrode to measure brain activity
Device: magnetoencephalogram — Implanting electrode to measure brain activity

SUMMARY:
Presurgical evaluation of epileptic patients require a precise mapping of cerebral regions implied in epileptic discharges and in normal function.

The current practice in most cases is to implant intracerebral electrodes in order to localize these regions in a reliable manner. However, non-invasive methods have been developed in order to record brain activity with no risk for the patient.

Still, it is necessary to validate and improve the signal processing methods and the underlying models these methods in order to optimize their use in clinical practice. To do so, it is necessary to record simultaneously electroencephalogram (EEG) and magnetoencephalogram (MEG) and stereo encephalogram SEEG (intracerebral). Such simultaneous recordings will permit to confront the exact same activity recorded non-invasively at the surface of the head, and represented on the brain thanks to the model and directly within the brain.

The objective is to define the conditions under which one can represent faithfully the activity measured intracerebrally from the surface measurements.

It will be record simultaneously MEG, scalp EEG and intracerebral EEG on a series of 60 patients. It will be record resting state signals, as well as stimulation protocols. The interictal epileptic discharges will be marked on the different modalities, and evoked potentials/fields computed in response to protocols. Sensitivity of recordings to activity visible on depth recordings will be evaluated as a function of localization of brain generators. Advanced signal processing methods will be used such as source localization and independent component analysis, in order to increase sensitivity of measures.

ELIGIBILITY:
Inclusion Criteria:

- Patients for whom implanting intracerebral electrodes is underway

Exclusion Criteria:

* Patients minors
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The number of epileptic discharges | 60 months
  Measurement of epileptic activity by electroencephalogram

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No